CLINICAL TRIAL: NCT05437562
Title: Pilot Investigation of Ewing Amputation in Veterans With Peripheral Arterial Disease Undergoing Below Knee Amputation
Brief Title: Randomized Clinical Trial for Ewing Amputation in the VA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SURG-001-21F; CX002366-01A1 (Other Grant/Funding Number: VA CSR&D Merit Award)
Record Dates: First submitted 2022-06-14; First posted 2022-06-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Peripheral Arterial Disease
Keywords: amputation
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: This study is evaluating an intervention in surgical technique for below knee amputation. The Veterans will be randomized to either Ewing amputation, which is a nuanced approach that incorporates RPNI and AMI to the standard below knee amputation. The standard below knee amputation is the comparison technique.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ewing Amputation (Experimental): Ewing Below Knee Amputation - incorporates RPNI and AMI
  Interventions: Procedure: Ewing Below Knee Amputation
- Standard Below Knee Amputation (Experimental): Standard Below Knee Amputation
  Interventions: Procedure: Standard Below Knee Amputation

INTERVENTIONS:
Procedure: Ewing Below Knee Amputation — Ewing Below Knee Amputation - incorporates RPNI and AMI
  Arms: Ewing Amputation
Procedure: Standard Below Knee Amputation — Standard Below Knee Amputation
  Arms: Standard Below Knee Amputation

SUMMARY:
This study follows the Pilot Investigation of Ewing Amputation for Veterans with PAD Undergoing a Below Knee Amputation. The 2 year pilot feasibility phase has concluded recruitment and enrollment.

The current phase is a 5 year randomized study of Ewing Below Knee Amputation vs. Standard Below Knee Amputation. If Veterans participate, they will be randomized to either Ewing Amputation or Standard Below Knee Amputation.

The scientific premise motivating this proposal is that Ewing Amputation is a promising surgical technique that may improve walking metrics in dysvascular Veterans by providing a better residual limb and improving pain and balance.

In preparation of this proposal, we have formed multi-disciplinary surgical teams at each site, and we have been supported by a clinical trial planning meeting to garner the considerable expertise in rehabilitation and amputee assessment from VA and DOD experts to assist in the design of this proposal, testing the overall hypothesis that: Ewing Amputation can help Veterans walk.

DETAILED DESCRIPTION:
Major amputations lead to significant challenges for Veterans and their loved ones. Thus, amputations and the care of amputees are a major focus of the VHA. Hence, the tripartite goals of the VHA Amputation System of Care (ASoC) are to: provide state of the art care, maximize health and independence, and to be the provider of choice for amputated Veterans. Veterans undergo ~1000 transtibial amputations (TTA) annually, making TTA a commonly performed operation in the VA. Almost all Veterans requiring TTA are dysvascular with peripheral artery disease (PAD) and/or diabetes. TTA is a safe operation with a low 30-day mortality rate, and ambulation with prosthesis rates are much better for TTA versus transfemoral amputations (TFA). Since ~50% of Veterans are satisfied with their ambulation after major amputation, improving ambulation is an important benchmark forward in the care of Veterans. Importantly, the lower ambulation rates in Veterans are attributed to modifiable sequelae of major amputation, including: slower wound healing9,10; chronic pain, imbalance, and falls. Excitingly, new techniques can improve pain and balance and may improve wound healing/prevent falls. Ewing amputation (EA) recreates the agonist-antagonist myoneural interface (AMI) maintaining muscle tension, proprioception and limiting fibrofatty muscle degeneration of muscle flaps. EA also creates regenerative peripheral neural interfaces (RPNI) to improve pain control. Thus, EA may have a significant benefit to Veterans undergoing TTA.

ELIGIBILITY:
Inclusion Criteria:

* Veterans who have reasonable blood flow to heal a TTA (defined as palpable popliteal pulse or palpable femoral pulse with popliteal artery signal)
* Veterans with an expectation of participating in rehabilitation and resuming ambulation after amputation (defined by the Veteran interest, recent ambulation by the Veteran, ability to participate in physical therapy as deemed by the investigators' physical therapy team)
* Veterans who will be undergoing below knee amputation for reasons other than infection (uninfected patients) or Veterans who have had foot infection localized below the ankle (retinaculum uninfected) that has been adequately debrided and treated with appropriate antibiotic course.

Exclusion Criteria:

* Veterans with end-stage renal disease (ESRD)
* Veterans requiring major amputation due to infection that includes the ankle retinaculum
* Veterans deemed to have inadequate blood flow to heal a TTA
* Veterans who cannot participate in rehabilitation or are not expected to be able to ambulate with a prosthesis for any reason
* Veterans who were randomized for their other limb (to prevent Veteran from the possibility of having 2 different amputations)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2030-02-02 (Estimated); Study Completion 2030-02-02 (Estimated)

PRIMARY OUTCOMES:
PROMIS Numeric Rating Scale | 12 months
  Patient reported rating scale to assess pain intensity and pain interference.
Socket Comfort Score | 12 months
  Patient reported rating scale to assess socket fit of prosthesis.
Phantom and Residual Limb Questionnaire | 12 months
  Patient reported questionnaire to assess sensation in phantom limb.
Lower Extremity Amputee Data Collection Form | 12 months
  Patient reported questionnaire to assess amputation system of care.
Lower Limb Mobility Rating Scale | 12 months
  Patient reported scale to assess movement with prosthetic leg.
Amputee Single Item Mobility Measure | 12 months
  Patient reported measure to assess current level of mobility.
Activities-specific Balance Scale | 12 months
  Patient reported scale to assess balance while performing every day activities.
Self-Reported Falls Measure | 12 months
  Patient reported one question survey to calculate falls in the previous month.
RAND Health Survey | 12 months
  Patient reported survey to assess general health while performing usual activities.
CRIS Fixed Form Instrument | 12 months
  Patient reported rating scale to assess usual activities in previous two weeks.
Patient Two Minute Walk Test | 12 months
  To measure distance patient can walk without assistance in 2 minutes.
Patient Timed Up and Go Test | 12 months
  To measure amount of time patient walks 3 meters.
Berg Balance Scale | 12 months
  To assess the patient's sitting and standing balance levels.
Amputee Mobility Predictor Questionnaire | 12 months
  To measure the patient's sitting, standing, turning and walking/stepping with and without prosthesis.

CONTACTS AND LOCATIONS:
Overall Officials: Luke P Brewster, MD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (3):
- United States (3):
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

IPD SHARING:
Plan to Share IPD: No